CLINICAL TRIAL: NCT01161199
Title: The Use of Leukapheresis to Support HIV Pathogenesis Studies
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: H52899-34904-01
Record Dates: First submitted 2010-07-09; First posted 2010-07-13 (Estimated); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: HIV
Keywords: HIV; latent reservoir; functional cure; leukapheresis
MeSH Terms: interventions — Leukapheresis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — CD4+ T cells Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Untreated non-controllers
  Interventions: Procedure: Leukapheresis
- Elite controllers
  Interventions: Procedure: Leukapheresis
- HAART-suppressed
  Interventions: Procedure: Leukapheresis

INTERVENTIONS:
Procedure: Leukapheresis — Blood will be taken by a needle placed in one arm and processed through a machine, which spins the blood so that the white blood cells will be separated out in the machine for purposes of this research and the rest of the blood will be returned through a needle in the other arm.

SUMMARY:
Despite the dramatic improvements that have resulted from combination antiretroviral treatment, long-term efficacy, toxicity, cost, and the requirements for life-long adherence remain as formidable challenges. Also, there is emerging consensus that persistent HIV-associated disease occurs during long-term highly active antiretroviral therapy (HAART). This disease may be due to either direct drug-toxicity and/or persistent viral replication/production and/or persistent HIV-associated inflammation. Hence, strategies aimed at achieving complete viral eradication may be needed in order to fully restore health among HIV infected individuals. Even if complete eradication proves impossible-as most believe to be the case-a less rigorous but still desirable outcome might be achieving durable control of virus in the absence of therapy. That a "functional" cure is possible is well illustrated by those rare individuals who are able to durably control replication competent virus in the absence of therapy ("elite" controllers).

A more complete understanding of the relationship between inflammation and viral persistence is necessary before more rationale studies of HIV eradication can be designed. Also, a well validated high through-put virologic assay needs to be developed that can estimate the size of the latent reservoir. Since the level of replication competent virus in long-term treated patients (and in elite controllers) is very small (< 1% of CD4 cells harbor HIV), large numbers of CD4+ T cells most be obtained from study participants in order to routinely isolate and quantify virus persistence.

ELIGIBILITY:
Inclusion Criteria:

* HIV seropositive
* Able to give informed consent
* Willing to undergo blood sampling and/or leukapheresis
* Meeting one of the following criteria: (1) on stable highly active antiretroviral therapy (HAART) with a recent undetectable viral load (< 50 copies/mL) ("HAART suppressed"), (2) antiretroviral untreated with an undetectable viral load (< 50 copies/mL) ("elite" controllers) and (3) antiretroviral untreated with a detectable viral load (> 1000 copies/mL) ("non-controllers")

Exclusion Criteria:

* Known anemia (HIV+ males Hct<34; females Hct<32) or contraindication to donating blood
* Blood coagulation disorder (including bleeding tendency or problems in past with blood clots)
* Platelets < 50,000/mm3
* PTT > 2x ULN
* INR > 1.5
* Albumin < 2.0 g/dL
* ALT > 5x ULN
* AST > 5x ULN
* Biopsy-proven or clinical diagnosis of cirrhosis
* Weight <120 lb
* High blood pressure > 160/100
* Low blood pressure < 100/70
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected patients on long-term antiretroviral therapy, untreated patients, and elite controllers will be studied.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-10-26 (Actual); Primary Completion 2033-07 (Estimated); Study Completion 2033-07 (Estimated)

PRIMARY OUTCOMES:
HIV DNA and RNA | Baseline and 6-12 months

CONTACTS AND LOCATIONS:
Overall Officials: Steven Deeks, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No